CLINICAL TRIAL: NCT01979835
Title: GYNEFIX-VIZ*: A STUDY OF SEROSAL-ANCHOR (SA) DISTANCE IN WOMEN IMMEDIATELY AND 6-8 WEEKS FOLLOWING INSERTION
Brief Title: GyneFix-Viz*: A Study of Serosal-Anchor (SA) Distance
Acronym: GF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wiebe, Ellen, M.D. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 130717
Record Dates: First submitted 2013-10-26; First posted 2013-11-08 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Contraception
Keywords: intrauterine device, contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GF (Experimental): Women who have a GyneFix Viz inserted
  Interventions: Device: GyneFix Viz

INTERVENTIONS:
Device: GyneFix Viz — insertion of GyneFix Viz and measurment of the SA distance

SUMMARY:
The GyneFix-Viz is a frameless copper intrauterine device (IUD) used for contraception. The GyneFix IUD has been marketed in Europe and Asia for about 10 years. The new anchor in the GyneFix IUD was designed to be more visible on ultrasound and this could improve safety by reducing failed insertions and perforations. We now need to know how easy it is for doctors to see and measure the distance of the anchor to the outside of the uterus. The purpose of this open, prospective, observational study is to assess the feasibility of measuring the distance from the serosa of the uterus to the anchor following insertion of the GyneFix-Viz and at follow-up 6-8 weeks later. Secondary objectives are to assess the ease and pain of insertion, the acceptability of the device to Canadian women and any complications. We will also compare expulsion rates in post-abortion and other women.

ELIGIBILITY:
Inclusion Criteria:

1. healthy women requesting intrauterine contraception
2. willing to have a GyneFix IUD for pregnancy prevention
3. able to return for a follow-up ultrasound
4. able to read and understand consent form

Exclusion Criteria:

1. Any contraindications precluding insertion of an IUD (e.g., infection, cancer of the uterus, malformation etc.)
2. Immediately after a pregnancy interruption > 10 weeks gestation

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1030 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R WIEBE, MD, Principal Investigator — University of BC
Locations (1):
- Willow Women's Clinic, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Women Who Enrolled to Have a GyneFix Viz Inserted: GyneFix Viz: insertion of GyneFix Viz and measurment of the SA distance
Period: Primary Outcome SA Measurment
Arm/Group | Women Who Enrolled to Have a GyneFix Viz Inserted
Started | 1030
Completed | 1012
Not Completed | 18
Not completed — failed insertion | 18
Period: Follow-up
Arm/Group | Women Who Enrolled to Have a GyneFix Viz Inserted
Started | 1012
Completed | 980
Not Completed | 32
Not completed — Lost to Follow-up | 32

BASELINE CHARACTERISTICS:
Groups:
- Women Enrolled to Have GF Inserted: All women requesting a GF and eligible for insertion who signed the informed consent document.
Arm/Group | Women Enrolled to Have GF Inserted
Number analyzed (Participants) | 1030
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1030
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1030

OUTCOME MEASURES:

1. Primary Outcome: Serosal-anchor Measurement
Description: endovaginal ultrasound measurement of the distance from the anchor of the device and the serosal surface of the uterus
Time Frame: 6-8 weeks
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Women Who Have a GyneFix Viz Inserted: GyneFix Viz: insertion of GyneFix Viz and measurment of the SA distance
Arm/Group | Women Who Have a GyneFix Viz Inserted
Number analyzed (Participants) | 1012
mm | 6.2 (2.7)

2. Secondary Outcome: Complications
Description: Number of participants with complications and removals at the end of the 5-year follow-up period
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Women Who Have a GyneFix Viz Inserted
Number analyzed (Participants) | 1012
Participants
  Perforation | 9
  Explusion | 36
  Pregnancy | 11
  Removed to conceive | 97
  Removed because no longer needed | 19
  Removed because >5 years | 95
  Removed due to symptoms and other reasons | 150
  Removed, missing reason | 83
  GyneFix in place | 420
  Missing | 92

ADVERSE EVENTS:
Arm/Group | Women Who Have a GyneFix Viz Inserted
All-Cause Mortality (participants affected / at risk) | 0/1012
Serious Adverse Events (participants affected / at risk) | 9/1012
Other Adverse Events (participants affected / at risk) | 180/1012
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Who Have a GyneFix Viz Inserted (N=1012)
perforation (Reproductive system and breast disorders) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Who Have a GyneFix Viz Inserted (N=1012)
expulsion (Reproductive system and breast disorders) | 36 (36) — IUD expulsion
pregnancy (Reproductive system and breast disorders) | 11 (11)
too much bleeding (Reproductive system and breast disorders) | 92 (92)
too much pain (Reproductive system and breast disorders) | 27 (27)
vaginal discharge (Reproductive system and breast disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No